CLINICAL TRIAL: NCT03945253
Title: A Phase 1, Open Label Study of ASP8374, an Immune Checkpoint Inhibitor, in Japanese Patients With Advanced Solid Tumors
Brief Title: Study of ASP8374, an Immune Checkpoint Inhibitor, in Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8374-CL-0102
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors
Keywords: Pharmacokinetics; Tumors; Oncology; Safety and tolerability; Locally advanced or metastatic solid tumor; ASP8374
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP8374-dose A (Experimental): Participants will receive dose A of ASP8374 solution intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP8374
- ASP8374-dose B (Experimental): Participants will receive dose B of ASP8374 solution intravenously on day 1 of every 3-week cycle.
  Interventions: Drug: ASP8374

INTERVENTIONS:
Drug: ASP8374 — Intravenous

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety profile and to characterize the pharmacokinetic profile of ASP8374 in Japanese patients with locally advanced (unresectable) or metastatic solid tumors.

This study also evaluates the anti-tumor effect of ASP8374.

DETAILED DESCRIPTION:
This study consists of two arms (Arm A: ASP8374 dose A; and Arm B: ASP8374 dose B). Arm B would only be opened if Arm A is deemed tolerable.

The study consists of 2 periods: Screening (up to 28 days) and treatment period. The Dose Limiting Toxicities (DLT) observation period is set at the beginning of the treatment period. A subject can continue to participate in the study after the end of the DLT observation period until discontinuation criteria are met. After discontinuation of study drug treatment, all subjects will complete an end of treatment visit and safety follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) that is confirmed by available pathology records or current biopsy and has received all standard therapies (unless the therapy is contraindicated or intolerable) felt to provide clinical benefit for his/her specific tumor type.
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Subject's last dose of prior antineoplastic therapy, including any immunotherapy, was at least 21 days prior to initiation of study drug administration. A subject with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) mutation-positive non-small cell lung cancer (NSCLC) is allowed to remain on EGFR tyrosine kinase inhibitor (TKI) or ALK inhibitor therapy until 4 days prior to initiation of study drug administration.
* Subject has completed any radiotherapy (including stereotactic radiosurgery) at least 2 weeks prior to initiation of study drug administration.
* Subject's adverse events (excluding alopecia) from prior therapy have improved to grade 1 or baseline within 14 days prior to initiation of study drug administration.
* Subject with metastatic castration resistant prostate cancer (mCRPC) (positive bone scan and/or soft tissue disease documented by computed tomography (CT)/ magnetic resonance imaging (MRI)) meets both of the following:

  * Subject has serum testosterone ≤ 50 ng/dL at screening.
  * Subject has had an orchiectomy or plans to continue androgen deprivation therapy (ADT) for the duration of study treatment.
* Subject has adequate organ function prior to initiation of study drug administration per specified laboratory values criteria within 7 days prior to initiation of study drug administration. If a subject has received a recent blood transfusion, the laboratory tests must be obtained ≥ 4 weeks after any blood transfusion.
* A female subject is eligible to participate if she is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 6 months after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the treatment period, and for 6 months after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the treatment period, and for 6 months after the final study drug administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner(s)) must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the treatment period, and for 6 months after the final study drug administration.
* Male subject with a pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the treatment period and for 6 months after the final study drug administration.
* Subject agrees not to participate in another interventional study while receiving study drug in present study (subjects who are currently in the follow-up period of an interventional clinical study are allowed).

Exclusion Criteria:

* Subject weighs < 45 kg at screening.
* Subject has received investigational therapy within 21 days prior to initiation of study drug administration. (A subject with EGFR activating mutations or a subject with an ALK mutation is allowed to remain on an investigational EGFR TKI or ALK inhibitor until 4 days prior to initiation of study drug administration.)
* Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to initiation of study drug administration. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone) are allowed.
* Subject has symptomatic central nervous system (CNS) metastases or subject has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Subjects with previously treated CNS metastases are eligible, if they are clinically stable and have no evidence of CNS progression by imaging for at least 4 weeks prior to initiation of study drug administration and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone or > 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Subject has an active autoimmune disease. Subjects with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy, or skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment are allowed.
* Subject was discontinued from prior immunomodulatory therapy due to a grade ≥ 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Subject has known history of serious hypersensitivity reaction to a known ingredient of ASP8374 or severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Subject has a known history of Human Immunodeficiency Virus.
* Subject is positive for Hepatitis B virus (HBV) antibodies and surface antigen (including acute HBV or chronic HBV) or Hepatitis C virus ([HCV] ribonucleic acid [RNA]). HVC RNA testing is not required in subjects with negative Hepatitis C antibody testing. HBV antibodies are not required in subjects with negative Hepatitis B surface antigen (HBsAg).
* Subject has received a live vaccine against infectious diseases within 28 days prior to initiation of study drug administration.
* Subject has a history of drug-induced pneumonitis (interstitial lung disease) or currently has pneumonitis.
* Subject has an infection requiring systemic therapy within 14 days prior to initiation of study drug administration.
* Subject has received a prior allogeneic bone marrow or solid organ transplant.
* Subject is expected to require another form of antineoplastic therapy while on study treatment.
* Subject has had a myocardial infarction or unstable angina within 6 months prior to initiation of study drug administration or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has had a major surgical procedure and has not completely recovered within 28 days prior to initiation of drug administration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by Dose Limiting Toxicity (DLT) | Up to 21 days
  DLT is graded using National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI-CTCAE] Version 4.03. The DLT observation period may be increased if deemed appropriate by the Tolerability Evaluation Meeting.
Safety and tolerability assessed by adverse events (AEs) | Up to 30 days after the last dose of study drug or until initiation of a new anti-cancer treatment, whichever comes first (a maximum of 109 weeks)
  An AE is any untoward medical occurrence in a subject administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Safety and tolerability assessed by immune-related AEs (irAEs) | Up to 30 days after the last dose of study drug or until initiation of a new anti-cancer treatment, whichever comes first (a maximum of 109 weeks)
  Most frequent immune-related AEs observed with currently approved checkpoint inhibitors include rash, oral mucositis, dry mouth, colitis/diarrhea, hepatitis, pneumonitis, and endocrinopathies .
Safety and tolerability assessed by serious adverse events (SAEs) | Up to 90 days after the last dose of study drug or until initiation of a new anti-cancer treatment, whichever comes first (a maximum of 117 weeks)
  An AE is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, life-threatening, persistent or significant disability/incapacity or substantial disruption, congenital anomaly or birth defect, hospitalization, or medically important event
Number of participants with laboratory value abnormalities and/or adverse events related to treatment | Up to 30 days after the last dose of study drug (a maximum of 109 weeks)
  Number of patients with potentially clinically significant laboratory values.
Safety and tolerability assessed by 12-lead electrocardiogram (ECG) | Up to end of treatment period (a maximum of 105 weeks)
  ECGs should be obtained after the subject has rested quietly and is awake in a fully supine position (or semi-recumbent, if supine is not tolerated) for 10 minutes before the first ECG from a triplicate or single ECG. Any clinically significant adverse changes on the ECS will be reported as (serious) AEs.
Number of participants with vital signs abnormalities and/or adverse events related to treatment | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  Number of patients with potentially clinically significant vital sign values.
Number of participants with physical exam abnormalities and/or adverse events related to treatment | Up to end of treatment period (a maximum of 105 weeks)
  Number of patients with potentially clinically significant physical exam values.
Safety and tolerability assessed by eastern cooperative oncology group (ECOG) performance status | Up to 30 days after the last dose of study drug (a maximum of 109 weeks)
  The ECOG Scale [Oken, 1982] will be used to assess performance status ; 0=Fully active, able to carry on all predisease performance without restriction; 1=Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, (e.g., light housework, office work); 2=Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
Pharmacokinetics (PK) of ASP8374 in serum: AUClast | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  AUClast: area under the concentration-time curve from the time of dosing up to the last measurable concentration. AUClast will be derived from the PK serum samples collected.
PK of ASP8374 in serum: AUCinf | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  AUCinf: AUC from the time of dosing extrapolated to time infinity. AUCinf will be derived from the PK serum samples collected.
PK of ASP8374 in serum: AUCinf(%extrap) | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  AUCinf(%extrap): Percentage of AUCinf due to extrapolation from the last measurable concentration to time infinity
PK of ASP8374 in serum: AUCtau | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  AUCtau: AUC from the time of dosing to the start of the next dosing interval at multiple dose conditions. AUCtau will be derived from the PK serum samples collected.
PK of ASP8374 in serum: Cmax | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  Cmax: maximum concentration. Cmax will be derived from the PK serum samples collected.
PK of ASP8374 in serum: Ctrough | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  Ctrough: trough concentration. Ctrough will be derived from the PK serum samples collected.
PK of ASP8374 in serum: tmax | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  tmax: time of maximum concentration. Tmax will be derived from the PK serum samples collected.
PK of ASP8374 in serum: t1/2 | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  t1/2: terminal elimination half-life. t1/2 will be derived from the PK serum samples collected.
PK of ASP8374 in serum: tlast | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  tlast: time of last measurable concentration. tlast will be derived from the PK serum samples collected.
PK of ASP8374 in serum: CL | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  CL: total clearance after intravenous dosing. CL will be derived from the PK serum samples collected.
PK of ASP8374 in serum: Vz | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  Vz: volume of distribution after intravenous dosing during the terminal elimination phase. will be derived from the PK serum samples collected. Vz will be derived from the PK serum samples collected.
PK of ASP8374 in serum: Vss | Up to 90 days after the last dose of study drug (a maximum of 117 weeks)
  Vss: volume of distribution at steady state after intravenous dosing. Vss will be derived from the PK serum samples collected.

SECONDARY OUTCOMES:
Percent change in tumor size from baseline | Up to end of treatment period (a maximum of 105 weeks)
  Tumor size is defined as the sum of the diameters of all target lesions per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The percent change from baseline in tumor size will be calculated for subjects with target lesions at baseline.
Best overall response (BOR) per RECIST 1.1 and 'immune' Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to end of treatment period (a maximum of 105 weeks)
  BOR is defined as the best response recorded from the start of the study treatment until the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP81001, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=406